CLINICAL TRIAL: NCT04061174
Title: A Comparison of the Effects of Shoulder Stabilization Exercises in Addition to Office Exercises on Scapular Dyskinesis, Muscle Strength, Posture and Proprioceptive Sensory Parameters in the Office Workers With Shoulder Protraction
Brief Title: Effects of Shoulder Stabilization Exercises in the Office Workers With Shoulder Protraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özde Depreli, Asst. Prof. Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODepreli
Record Dates: First submitted 2019-07-26; First posted 2019-08-19 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Work-Related Condition
Keywords: shoulder; proprioception; vibration; posture; stabilization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder stabilization exercise and office exercise training (Experimental): Shoulder stabilization exercises will be given to the experimental group participants individually during 8 weeks. Exercises will be done 3 times a week and each exercise will be performed with 10 repetitions, 3 sets and 60-90 seconds rest between sets. Also experimental group participants will do office exercise training that given to other group participants.
  Interventions: Other: Shoulder stabilization exercises
- Office exercise training (Experimental): Office-based stretching exercises will be given to other group 3 sets will be applied by waiting 15 seconds for increasing range of motion of back, shoulder and neck joints.
  In addition, isometric exercises and scapula stabilization exercises will be given to strengthen the shoulder muscles and participants will do these exercises 3 times a week and once a day in 10 repetitions (10-15 seconds) and 3 sets. Each set will be given a rest of 60-90 seconds. Total time will be 10-15 minutes.Office exercise training will last a total of 8 weeks.
  Interventions: Other: Office exercises training

INTERVENTIONS:
Other: Shoulder stabilization exercises — When participants are able to do the exercise 15 repetitions without difficulty, the exercise will be advanced by modifying or adding the weight.The exercises include chin tulk exercise, shoulder closed chain weight transfer, prone and iso-abdominal exercises, push-up exercise, lower trapezius muscle strengthening exercise, dead bug exercise, ball rolling on the wall, bench press with dumbbell and internal/external rotation (IR / ER) strengthening exercises
  Other Names: Shoulder stabilization exercises and office exercises training
  Arms: Shoulder stabilization exercise and office exercise training
Other: Office exercises training — Information will be given in a brochure that includes the appropriate chair height and work table, sitting position, distance between eyes and monitor, and table chair dimensions.approved and standardized office-based stretching and strengthening exercises will be given for workplaces
  Arms: Office exercise training

SUMMARY:
Office workers continuously work with the forward head posture. Forward head posture may cause upper extremity problems in the office workers due to the increase in the load on the muscles and joints of the cervical spine. This working posture may cause scapular rotation downward, increase in activation of the scapular muscles, pain, limited range of motion (ROM) and poor proprioception, which can create a vicious circle. Especially in the office workers that using computer vibration sensation reduction and upper extremity problems are seen. The aim of this study is to investigate the effect of shoulder stabilization exercises on scapular dyskinesis, muscle strength, posture and proprioceptive sensory parameters in addition to office exercises in the office workers with shoulder protraction.

DETAILED DESCRIPTION:
The study is planned so that scapular dyskinesia, muscle strength, posture and proprioceptive sense measurements will be taken at 3 different times (before treatment, 8th week and 12th week) for two independent groups (control and experimental groups).Based on the proprioception sense findings in our previous pilot study, the intergroup effect size was predicted to be approximately 0.35 (weak to moderate). Assuming that type I error is 5%, type II is 20%, and the correlation between repeated measurements is 80% (high correlation), the total sample size obtained with the help of G Power 3.1.9.2 software is calculated as 60 people. Individuals are randomly divided into two groups (by blocking method). Groups are matched by stratified random sampling/proportionate distribution by degree of shoulder protraction (acromion level below and above 6.5 cm) and gender.

Study data will be analyzed using the statistical software [Statistical Package For The Social Sciences Software (SPSS 25.0)].Frequency and percentage for continuous data, mean, standard deviation, minimum and maximum value for categorical data will be reported. Independent sample t-test to determine the difference according to the groups in continuous variables, analysis of variance in repeated measures to determine the change over time, two-way analysis of variance in repeated measures with repetitions on a single factor to evaluate the group and time change together. Pearson chi-square and Fisher-Freeman-Halton test will be performed model to evaluate the difference according to groups in categorical variables. Bonferonni correction will be used for multiple comparisons, Friedman S and Cochran Q tests will be used to evaluate time-dependent variation, and two-way analysis of variance will be used for repeated measures with repetitions on a single factor to evaluate group and time variation together.The significance level will be accepted as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 25-40 age range
* Participants that working at the desk for at least 1 year and more than 4 hours per day
* Participants with The Disabilities of the Arm, Shoulder and Hand Score of 15 or less
* Participants with pain severity of neck and upper extremity is 2 cm or less on visual analog scale in the last 6 months

Exclusion Criteria:

* Participants with disc herniation, spondylisthesis, degenerative arthritis or related surgery
* Participants with rotator cuff injury, acromioclavicular separation, dislocation and related surgical operations
* Participants with problems such as diabetes, rheumatoid arthritis, ankylosing spondylitis, severe osteoarthritis
* Participants who have received physiotherapy for the neck and upper extremity in the last 6 months

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of shoulder proprioception sense | 15 minute
  Evaluation of shoulder proprioception will be performed with an isokinetic (Cybex Norm) dynamometer that is found as the most reliable method of shoulder proprioception measurement.Functionally, a proprioceptive testing device (PTD) will be used to measure kinesthesia as the threshold to detect passive motion and measure joint position sense by the ability to reproduction of passive positioning and reproduction of active positioning
Assessment of shoulder vibration sense | 5 minute
  Shoulder vibration sense evaluation will be performed with Vibrometer (Diabetic Foot Care, India), which has demonstrated high reproducibility and reliability.

SECONDARY OUTCOMES:
Rapid upper limb assessment (RULA) tool | 5 minute
  Ergonomic risk factors will be determined through direct observation of employees' postures by the dominant side in their workplace using the RULA tool. RULA assesses biomechanical and postural loading on the upper limbs. It is divided into two segments (A and B). Segment A includes steps regarding the assessment of upper arm, lower arm and wrist, whereas segment B is related with the assessment of neck, trunk and legs. Zero and 1 points were added to A and B scores by depending on the muscle use (static postures held for longer than one minute or repeated more than four times per minute) and force (total hours of work in a day) and consequently C and D scores were achieved. Then, C and D scores were combined in a table to obtain a Grand Score. The grand score ranges from 1 to 7 in which a score of 1 or 2 is acceptable, a score of 3 or 4 needs further investigation, 5 or 6 needs investigation and changes sooner and a score of 7 needs immediate investigation and change.
Pectoralis minor length measurement | 2 minute
  Participants will be instructed to stand in a normal, relaxed posture during data collection. The examiner palpate the medial-inferior angle of the coracoid process of the scapula and just lateral to the sternocostal junction of the inferior aspect of the fourth rib and measured the distance between these landmarks with caliper. Three measurements will be taken; the average is divided by the participant's height and multiplied by 100 to calculate the pectoralis minor length index for analysis
Passive internal rotation (IR) and external rotation (ER) mobility flexibility | 5 minute
  Using standard goniometer techniques, passive shoulder IR and ER with the subject supine and the arm abducted 90˚, elbow flexed to 90 ˚and the forearm in neutral rotation. Passive ER will be measured by moving the subject's extremity into ER, maintaining positions of the abduction, elbow flexion and forearm rotation. The extremity will be rotated externally until end range of motion is obtained. To measure IR, the subject's arm is internally rotated while an anterior force will be applied to the coracoid and humerus to ensure that scapular compensation don't occur. All measurements will be taken three times, and a mean of the three measurements will be calculated in degree.
Active internal rotation (IR) and external rotation (ER) mobility flexibility | 5 minute
  Spinous process of the cervical 7 (C7) and thoracic 5 (T5) vertebra will be identified as reference points. The subject is standing with feet shoulder width apart. With thumb extended, the subject reached extremity upwards and towards the midline to a maximum hand behind back position. Tape measure will be used to record the distance in centimetres from the thumb tip to T5 spinous process for active IR mobility. Also subject will be asked to make maximum external rotation by moving harm behind neck with the thumb pointing down and the distance from thumb to C7 will be measured with tape measure for active ER mobility.
Muscle Strength Measurement | 40 minute
  Upper, middle and lower trapezius, anterior, middle and posterior deltoid, serratus anterior, supraspinatus, infraspinatus, latissimus dorsi and pectoralis major-minor muscle strength measurement will be performed by hand-held dynamometer.3 repetitions at 30 seconds intervals and the average value will be recorded.
Closed Kinetic Chain Upper Extremity Stability test | 5 minutes
  The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) is examining upper limb stability. It consists of counting how many times the subject performs alternating touches on the opposite hand in a closed kinetic chain position (push-up) over 15 seconds, with three trials. The normalized score is obtained by dividing the number of touches by subject height.
Passive glenohumeral (GH) horizontal adduction mobility flexibility | 5 minutes
  To assess GH horizontal adduction, subjects are positioned supine with both shoulders flush against a standard examination table. Shoulder and elbow is in 90˚ of both abduction and flexion. The tester's passively move the humerus into horizontal adduction. To measure GH horizontal adduction, the digital inclinometer is aligned with the ventral midline of the humerus. The angle is created by the end position of the humerus with respect to 0˚ of horizontal adduction (perpendicular plane to the examination table, as determined by the digital inclinometer) is then recorded as the total amount of GH horizontal adduction motion in degree.
Total scapula distance | 2 minutes
  The distance from the anterior aspect of the acromion to the T3 spinous process will be measured with a caliper while the subject is standing in a relaxed position. Distance will be recorded in cm
Scapula upward rotation measurement | 10 minutes
  All subjects will assessed in a relaxed, standing (barefoot) position and asked to perform full extension at the elbow, neutral wrist position, and with the thumb leading in the coronal plane. One inclinometer will be attached parallel to the humerus with use of a tape. Scapular upward rotation will be measured using the second inclinometer. Subjects are asked to actively move their arms (dominant or non-dominant randomly) from rest position to 45˚, from rest position to 90˚and from rest position to 135˚ abduction and to hold arm in these positions for measurement (measured with first inclinometer) in frontal plane (randomly). Three trials with a 30 s rest between trials wiil be performed for each shoulder (at rest position, 45˚, 90˚ and 135˚ abduction) and means of them will be calculated.
Lateral Scapular Slide Test (LSST) | 5 minutes
  LSST will be used for assessing scapular asymmetry under varying load positions. Measurements of scapular position are taken while scapular position with the arm abducted 0, 45, and 90 degrees in the coronal plane. Distance from the inferior angle of the scapula to the spinous process of the thoracic vertebra in the same horizontal plane will be measured in all 3 position. If the distance is greater than 1.5cm, it means LSST is positive.
Cervical posture analysis by photographing method | 10 minutes
  Tripod and camera (Canon Rebel T5i, 18.0 megapixel) will be located 0.8 meters away from the participant, at C7 alignment in a position, where the lens of the camera will be vertical to the individual's sagittal level. Reflective markers will be placed on the lateral canthus of the eye, the tragus of the ear, the spinous process of C7. The sagittal head angle will be formed at the intersection of a horizontal line through the tragus of the ear and a line joining the tragus of the ear and the lateral canthus of the eye. The cervical angle is highly reliable to assess the forward head position. It is the angle formed at the intersection of a horizontal line through the spinous process of C7 and a line to the tragus of the ear. Triangular screen ruler program will be used for calculate angles.
Sagittal shoulder posture analysis by photographing method | 10 minutes
  Tripod and camera (Canon Rebel T5i, 18.0 megapixel) will be located 0.8 meters away from the participant, at C7 alignment in a position, where the lens of the camera will be vertical to the individual's sagittal level. Reflective markers will be placed on the the spinous process of C7 and lateral shoulder. Where a horizontal line passing through the lateral shoulder meets the line drawn from C7 to the lateral shoulder, the point of intersection forms the sagittal shoulder-C7 angle. It indicates the degree of roundedness of the shoulders. A protracted shoulder would yield a lesser value of this angle. Triangular screen ruler program will be used for calculate angle.
Coronal shoulder posture analysis by photographing method | 10 minutes
  Tripod and camera (Canon Rebel T5i, 18.0 megapixel) will be located 0.8 meters away from the front of participant. Reflective markers will be placed on the left and right coracoid processes. It is defined as the angle between a horizontal line and a line joining the coracoid processes. It is used to determine whether the left and the right shoulders are level or not. Its normal value should be 180 degrees. Triangular screen ruler program will be used for calculate angle.
Thoracic posture analysis by photographing method | 10 minutes
  Tripod and camera (Canon Rebel T5i, 18.0 megapixel) will be located 0.8 meters away from the participant, at C7 alignment in a position, where the lens of the camera will be vertical to the individual's sagittal level. Reflective markers will be placed on the spinous process of C7 and the spinous process of thoracic 12 (T12). The point where lines (perpendicular to the skin surface) produced through T12 and C7 markers intersect each other forms the thoracic flexion angle. The lesser the value, the less is the kyphosis. Triangular screen ruler program will be used for calculate angle.

CONTACTS AND LOCATIONS:
Overall Officials: Ozde Depreli, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Mersin 10 Turkey, Cyprus

IPD SHARING:
Plan to Share IPD: No
When authors requesting results and contact me, I will share data results with them.